CLINICAL TRIAL: NCT02074072
Title: Comparison of Glidescope, Pentax-AWS and Macintosh Laryngoscope for Intubation During Chest Compression in 15-30 Degree Left-Lateral Tilt: A Manikin Simulation Study of Maternal Cardiopulmonary Resuscitation
Brief Title: Endotracheal Intubation Using Three Laryngoscopes in Maternal Cardiac Arrest: a Manikin Simulation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Lee Sang Hyun, clinical fellow, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HYI-14-004-1
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Cardiac Arrest
Keywords: Endotracheal intubation; Left lateral tilt wedge; Maternal Cardiopulmonary Resuscitation; Manikin Study
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Direct laryngoscope (Experimental): Macintosh laryngoscope
  Interventions: Device: 15 degree left-lateral tilt wedges; Device: 30 degree left-lateral tilt wedges
- Videolaryngoscope-1 (Experimental): Glidescope
  Interventions: Device: 15 degree left-lateral tilt wedges; Device: 30 degree left-lateral tilt wedges
- Videolaryngoscope-2 (Experimental): Airwayscope
  Interventions: Device: 15 degree left-lateral tilt wedges; Device: 30 degree left-lateral tilt wedges

INTERVENTIONS:
Device: 15 degree left-lateral tilt wedges — The wedges are made of aluminium
  Other Names: Custom-made hard wedges
Device: 30 degree left-lateral tilt wedges — The wedges are made of aluminium
  Other Names: Custom-made hard wedges

SUMMARY:
European Resuscitation Council (ERC) Guidelines for Resuscitation 2010 emphasize high quality chest compressions .They propose minor changes for pregnant women: manual left deviation of the uterus or a left-lateral incline of 15-30to alleviate pressure on the inferior vena cava. We will examine the performance of the Glidescope (GVL), the Pentax-AWS Airwayscope(AWS) and Macintosh laryngoscope (McL) for airway management during chest compressions on 15 and 30 degree left-lateral tilt (15 &30 LLT) custom-made hard wedges.

DETAILED DESCRIPTION:
Materials

1. Sim Mom manikin (Laerdal, Stavanger, Norway)
2. Stryker ST104-747(Transport stretcher®, 760 x 2110 mm, 228 kg, Stryker Co., Kalamazoo, Michigan, US)
3. LUCAS Chest Compression System( LUCAS Chest Compression System, Physio-Control/Jolife AB)
4. Backboard(450 ×600 ×10 mm, 3 kg Lifeline Plastic, Sung Shim Medical Co., Bucheon, Korea)

ELIGIBILITY:
Inclusion Criteria:

* Experience of intubation > 50 times
* Postgraduates year 1,2,3,4 and Emergency physicians in emergency department

Exclusion Criteria:

* Wrist or Low back disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Time to intubation | 1day
  We will check the times from inserting blade to mouth to exposing vocal cord and from exposing vocal cord to first ambu-bagging.
Success rate of intubation | 1day
  Definition of failed intubation
  * Time to intubation is longer than 90 seconds.
  * Wrong placement of endotracheal tube (For example : Esophageal intubation etc.)

SECONDARY OUTCOMES:
Laryngeal View during intubation | 1day
  We will record the best laryngeal View during intubation. We will record according to the Cormack-Lehane Grade system.
The preference for laryngoscopes | 1day
  1. The preference for laryngoscope regardless of tilting degree of wedges
  2. The preference for laryngoscope in 15 degree left-lateral tilt situation .
  3. The preference for laryngoscope in 30 degree left-lateral tilt situation . (Participants will select only 1 of 3 laryngoscopes and the preference will be displayed as histogram)

CONTACTS AND LOCATIONS:
Overall Officials: Sang hyun Lee, M.D, Principal Investigator — Hanyang University Seoul Hospital
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea